CLINICAL TRIAL: NCT00354406
Title: A Randomized Trial Comparing the Efficacy on Myocardial Infarct Size Reduction of Early vs. Late Abciximab Administration During Primary Percutaneous Coronary Angioplasty
Brief Title: Efficacy Study on Early Versus Late Abciximab Administration During Primary Coronary Angioplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pisa (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Prof. Anna Sonia Petronio, Head of Cardiac Catheterization Laboratory, University of Pisa, Azienda Ospedaliero-Universitaria Pisana, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP-DCT-200601
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Myocardial Infarction
Keywords: Abciximab; Magnetic Resonance Imaging; Percutaneous Transluminal Coronary Angioplasty
MeSH Terms: conditions — Myocardial Infarction | interventions — Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients in Arm A (Early abciximab arm) will receive abciximab at time of STEMI diagnosis, before transfer to the Cath Lab to undergo primary angioplasty.
  Interventions: Drug: abciximab
- B (Active Comparator): Patients in Arm B (Late abciximab arm) will receive abciximab at time of primary angioplasty, directly in the Cath Lab.
  Interventions: Drug: abciximab

INTERVENTIONS:
Drug: abciximab — standard i.v. bolus of abciximab is administered at time of randomization in arm A, and at time of primary angioplasty in arm B.

SUMMARY:
Abciximab has been demonstrated to improve outcome when administered during primary angioplasty in patients with acute myocardial infarction. The Primary Objective of the study is to demonstrate that early (before transportation form remote hospital to the cath lab) abciximab administration during acute myocardial infarction reduces infarct size as compared with late (just prior to PCI) abciximab administration, as measured by delayed enhancement magnetic resonance (MR) at 6 months.

DETAILED DESCRIPTION:
Strategies directed at improving myocardial perfusion or viability in the setting of acute myocardial infarction (AMI) are currently suboptimal. The consequences of microvascular damage, as assessed by the TIMI myocardial perfusion (TMP) grade or by cardiac magnetic resonance imaging (MR), are serious and affect survival after AMI. Because the size of the infarct is an important predictor of prognosis, precise determination of infarct size allows risk stratification of patients after AMI.

First-pass MR perfusion studies recently developed provide quantification of the absolute measure of myocardial blood flow as well as direct visualization of myocardial perfusion abnormalities, such as areas of "no-reflow". The hyperenhancement technique (Delayed enhancement) identifies viable and nonviable myocardium as well as no-reflow areas.

A recent pilot study showed that infarct size measured by scintigraphy at 7 days was 23% vs 14% when abciximab was administered in the cath lab vs emergency room, with a reduction in infarct size of 40%.

The present study will be conducted at the Cardiothoracic Department of the University of Pisa together with the Institute of Clinical Physiology (CNR) and two other Cath Labs of the West of Tuscany. Each Cath Lab will treat patients enrolled in peripheral hospitals referring the patients for primary PCI.

The primary objective of the study is to demonstrate that early abciximab administration (before transfer) as compared with late abciximab administration (in the Cath Lab) reduces infarct size as measured by delayed hyperenhancement imaging at 6 months.

The major secondary objectives of this substudy are to demonstrate that early abciximab administration:

1. Improves angiographic TMP grade and cTFC compared with primary PCI group, immediately after PCI.
2. Reduces the extension of no-reflow areas, as assessed by DE-MRI before discharge.
3. Reduces the extension of microvasculature damage as assessed by fist-pass perfusion study by MRI before discharge.
4. Improves regional wall motion and left ventricular ejection fraction (LVEF) as measured by cine MR and 2D echocardiography at 6 months
5. Reduces the occurrence of LV remodeling at 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Prolonged, continuous signs and symptoms of ischemia lasting more than 20 min, starting within 6 hours prior to randomization, and ST segment elevation ≥ 2mm or new left bundle branch block
* Absence of contraindications to Abciximab (for details cf. below section)
* Written informed consent

Exclusion Criteria:

* Low-risk (ST elevation in ≤2 leads) inferior AMI
* Previous infarction in the same area (assessed by ECG)
* PCI in the 2 weeks prior to AMI
* Know hypersensitivity to abciximab
* Active internal bleeding
* History of cerebrovascular accident in the previous 2 years or cerebrovascular accident with a significant residual neurological deficit
* Head or spine surgery or trauma in the previous 2 months
* Recent (within six weeks) gastrointestinal (GI) or genitourinary (GU) bleeding of clinical significance
* Administration of oral anticoagulants within seven days unless prothrombin time is <1.2 times control
* Bleeding diathesis or severe uncontrolled arterial hypertension
* Thrombocytopenia (<100 000 cells/mL)
* Recent (within six weeks) major surgery or trauma
* Intracranial neoplasm, arteriovenous malformation, or aneurysm
* Severe renal or liver failure
* Allergy to aspirin
* Contraindication to MRI examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
infarct size (% of left ventricular mass) as measured by delayed hyperenhancement magnetic resonance imaging at 6 months | at 6 months after myocardial infarction

SECONDARY OUTCOMES:
Angiographic TIMI Myocardial Perfusion grade and corrected TIMI frame count, assessed immediately after PCI. | final angiography at the end of PCI
Extension of no-reflow areas (% of left ventricular mass), as assessed by delayed enhancement-MRI before hospital discharge. | At day 4-5 after myocardial infarction.
Extension of microvasculature damage (% of left ventricular mass), as assessed by fist-pass perfusion study by MRI before hospital discharge. | At day 4-5 after myocardial infarction
Regional wall motion and left ventricular ejection fraction, as measured by cine MRI and 2D echocardiography at 6 months | at 6 months after myocardial infarction
Rate of left ventricular remodeling (increase in end-diastolic volume >20%), as measured by cine MRI and 2D echocardiography at 6 months | at 6 months after myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Petronio, MD, Principal Investigator — University of Pisa
Locations (1):
- Cardiothoracic Department, Ospedale Cisanello, Pisa, Italy

REFERENCES:
- [Background] Al-Saadi N, Nagel E, Gross M, Schnackenburg B, Paetsch I, Klein C, Fleck E. Improvement of myocardial perfusion reserve early after coronary intervention: assessment with cardiac magnetic resonance imaging. J Am Coll Cardiol. 2000 Nov 1;36(5):1557-64. doi: 10.1016/s0735-1097(00)00914-1. PMID 11079658